CLINICAL TRIAL: NCT03276897
Title: Efficacy and Tolerance Evaluation of a "Revitalizing" Face Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0517
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Face Aging/Photo Aging of Moderate Grade

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutriage SPF 30 day cream and Nutriage night cream (Experimental): Application of the study products (day cream at the morning and night cream at the evening), for an uninterrupted period of 3 months.
  Interventions: Other: Nutriage SPF 30 day cream and Nutriage night cream (Difa Cooper S.p.a, Italy)

INTERVENTIONS:
Other: Nutriage SPF 30 day cream and Nutriage night cream (Difa Cooper S.p.a, Italy) — A fixed quantity of both cosmetic products was applied for an uninterrupted period of 3 months, on the face included the submental area (day cream at the morning and the night cream at the evening), preferentially always at the same hour, with a mild massage

SUMMARY:
Efficacy and Tolerance Evaluation of a"revitalizing" face treatment consisting of a day and a night cream

DETAILED DESCRIPTION:
Aim of the study was to evaluate clinically and by non-invasive instrumental evaluations the activity of a "revitalizing" face treatment consisting of a day and a night cream, applied for an uninterrupted period of 3 months, by female volunteers, aged 35-60 years, with aging/photo aging of moderate grade.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* age 35-60 years,
* Caucasian subjects,
* presence of moderate face ritidosis,
* agreeing to present at each study visit without make-up,
* accepting to follow the instructions received by the investigator,
* accepting to not change their habits regarding food, physical activity, face cleansing and make- up use,
* agreeing not to apply or take any product or use face massages or other means known to improve skin wrinkle and skin qualities during the entire duration of the study,
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study,
* no participation in a similar study currently or during the previous 3 months
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Pregnancy,
* lactation,
* sensitivity to the test products or their ingredients (to be assessed by the investigator during the baseline visit),
* subjects whose insufficient adhesion to the study protocol is foreseeable.
* presence of cutaneous disease on the tested area as lesions, scars, malformations,
* recurrent facial/labial herpes,
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* endocrine disease,
* hepatic disorder,
* renal disorder,
* cardiac disorder,
* pulmonary disease,
* cancer,
* neurological or psychological disease,
* inflammatory/immunosuppressive disease,
* drug allergy.
* anti-inflammatory drugs, anti-histaminic, topic (application on the face) and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of hormonal treatment starting more than 1 year ago),
* using of drugs or dietary supplements able to influence the test results in the investigator opinion.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change of wrinkles grade, around the eyes (Crow's feet) | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Variation of wrinkles grade from baseline of the Glogau's reference photographic scale (visual score from 1-4) where:
  * Type 1: early wrinkles
  * Type 2: wrinkle in motion
  * Type 3: wrinkles at rest
  * Type 4: Only wrinkles
Change of wrinkles grade of nasolabial folds | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Variation of wrinkles grade from baseline of the Lemperle's reference photographic scale (visual score from 1-6) where:
  * Grade 1: no wrinkles
  * Grade 2: just perceptible wrinkles
  * Grade 3: shallow wrinkles
  * Grade 4: moderately deep wrinkles
  * Grade 5: deep wrinkles, well-defined folds
  * Grade 6: very deep wrinkles, redundant fold
Change of skin surface microrelief's regularity | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Variation of skin surface microrelief's regularity grade from baseline of cheek surface microrelief photographic scale where:
  * Grade 1:very regular
  * Grade 2: regular
  * Grade 3: irregular
  * Grade 4: very irregular.
Change of skin resistance to pinching clinical score | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  The evaluation was performed at level of cheek (malar region) according to the following score:
  0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Change of skin resistance to traction clinical score | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  The evaluation was performed at level of cheek (malar region) according to the following score:
  0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Change of skin recovery after pinching clinical score | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  The evaluation was performed at level of cheek (malar region) according to the following score:
  0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Change of skin dryness clinical score | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Clinical evaluation of skin dryness was performed according to the following score:
  0 = very hydrated skin
  1. = hydrated skin
  2. = normal skin
  3. = kindly dry skin
  4. = dry skin
  5. = very dry skin
Change of vascular and pigmentary homogeneity clinical score | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Homogeneity grade was determined according to specific reference clinical and photographic scales and to the following clinical score:
  0 = very homogeneous
  1. = homogeneous
  2. = quite not homogeneous
  3. = not homogeneous
  4. = very not homogeneous
  5. = marked not homogeneous

SECONDARY OUTCOMES:
Change of roughness profilometric parameters | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Crow's feet profilometric parameters measured by Primos compact portable device (GFMesstechnik). Ra is average roughness of the analysed profile, Rt is wrinkles total high, Rv is wrinkles maximum depth.
Photographic documentation (3D pictures) | Baseline visit (T0), 1 month (T1), 2 months (T2), 3 months (T3)
  Three-dimensional pictures of the face taken by VECTRA H1 handheld imaging system.

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Monza, Monza-brianza, Italy